CLINICAL TRIAL: NCT02403479
Title: Phase 2 Study Examining the Effects of Topical Intranasal Silver Colloid in Patients With Recalcitrant Chronic Rhinosinusitis
Brief Title: The Effectiveness of Topical Silver Colloid in Treating Patients With Recalcitrant Chronic Rhinosinusitis
Acronym: CRS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Leigh Sowerby, Assistant Professor, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 106309
Record Dates: First submitted 2015-03-01; First posted 2015-03-31 (Estimated); Results first posted 2019-11-15 (Actual); Last update posted 2019-11-15 (Actual); Status verified 2019-10

CONDITIONS: Rhinosinusitis
MeSH Terms: conditions — Rhinosinusitis | interventions — colloidal silver; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Saline then Silver Colloid (Experimental): Each participant uses 6 weeks of Saline first (Frequency= 2 sprays twice daily; Route= topical intra-nasal spray; Duration= 6 weeks) followed by 6 weeks of silver colloid (Dose= 6.7mcg silver daily; Frequency= 2 sprays twice daily; Route= Topical intra-nasal spray; Duration= 6 weeks)
  Interventions: Drug: Silver Colloid; Other: Saline
- Silver Colloid then Saline (Experimental): Each participant uses 6 weeks of Silver Colloid first (Dose= 6.7mcg silver daily; Frequency= 2 sprays twice daily; Route= Topical intra-nasal spray; Duration= 6 weeks) followed by 6 weeks of saline (Frequency= 2 sprays twice daily; Route= topical intra-nasal spray; Duration= 6 weeks).
  Interventions: Drug: Silver Colloid; Other: Saline

INTERVENTIONS:
Drug: Silver Colloid — Topical silver colloid will be administered for 6 weeks. This will either occur before topical saline nasal spray. Participants are randomized as to the order of sprays. The commercially available silver colloid product, Sovereign Silver Mineral Supplement, will be used.
  Other Names: Silver Hydrosyl by Sovereign Silver
Other: Saline — Topical saline will be administered for 6 weeks. This will occur before the topical silver colloidal nasal spray. Participants are randomized as to the order of sprays.

SUMMARY:
Chronic rhinosinusitis without polyposis (CRSsP) is a very common condition that occurs when the lining of the sinuses becomes persistently irritated. Standard management options include topical steroids, antibiotics and surgery, but treatment-resistant CRSsP is frequently encountered. Bacterial biofilms are routinely detected within the nasal mucosa of CRSsP patients and are now thought to play an important role in the protracted nature of the disease. Colloidal silver is a widely used naturopathic agent that has recently been shown to eliminate bacteria, and in particular in vitro sinusitis biofilms, in laboratory studies. Although silver is currently used in a variety of chronic wound therapies, it has not yet been formally studied in people with CRSsP. It is our intention with this project to determine whether colloidal silver is a useful treatment strategy for patients with refractory CRS.

DETAILED DESCRIPTION:
The paranasal sinuses are within the bones of the face and head. Six paired sinuses are present in humans, and although their exact function is a topic for debate, they appear to play several roles ranging from cushioning the brain during trauma to increasing resonance of the voice and releasing nitric oxide to help with lung physiology. The sinuses are lined with a layer of respiratory epithelium that normally secretes a small amount of mucus to keep the sinuses lubricated and contains cilia to help sweep away debris. Rhinosinusitis occurs when this lining gets infected or irritated which can lead to excessive mucus production and impaired mucus drainage. It is a very prevalent condition affecting up to 16% of the population and is the fifth most common diagnosis generating an antibiotic prescription1,2.

Chronic rhinosinusitis without polyposis (CRSsP) is characterized by persistent symptoms of nasal congestion, mucus discharge from the nose, facial pain or anosmia for at least three months. Unlike acute rhinosinusitis, which is usually caused by infection, CRSsP can have more elusive causes and can be profoundly more complicated.3 Due to the challenging nature of CRS, physicians often use a variety of treatment strategies against it.3 Potential treatments for CRSsP include lifestyle modifications (quitting smoking, reduce allergen exposure, etc.), nasal saline irrigations, nasal corticosteroid spray or irrigations, antibiotics and surgery. Typically, there is a stepwise fashion to the therapy offered to patients whereby the more aggressive or invasive modalities are reserved for those who did not benefit from simpler approaches. Even despite all these regimens there is a small subset of patients who continue to fare poorly. One thought toward the reason for this centers on the frequent presence of biofilms within the sinuses of recalcitrant CRSsP patients.4

Biofilms have been reported in CRS populations for a decade now by a number of authors.4,5 Furthermore, their presence has been linked to more severe disease both pre and post-operatively. Using fluorescence in situ hybridization investigators have been able to identify staphylococcus aureus (S. aureus) and Haemophilus influenza (H. influenza) as the most common biofilm-forming organisms.5 In fact, H. influenza biofilms seem to be more common in milder patterns of CRS, whereas S. aureus biofilms are present in more severe, refractory forms of the disease.5 A very recently published study demonstrated colloidal silver directly attenuating S. aureus biofilms in vitro and herein lays the premise of our study.6

Interest in colloidal silver, a commercially available naturopathic product, was sparked after clinical improvements were seen in a number of recalcitrant CRS patients who sprayed the agent intranasally. Silver has long been used for its bactericidal properties, as it is one of the most toxic elements to microorganisms.7 Silver-impregnated dressings and catheters are currently used in the treatment of burns, ulcers and chronic wounds. Clear advantages of silver over modern antibiotics include broad spectrum activity against Gram-positive and Gram-negative organisms, fungi, protozoa and some viruses as well as the general absence of resistance developing in a number of bacterial species.7,8 In addition, silver has been shown to have activity against Pseudomonas aeruginosa biofilm development.9

The main reasons colloidal silver fell out of use as an antiseptic are due in large part to the advent of antibiotics, uncertain safety, and the production of argyria on ingestion10. Although it is not yet known which dose of silver is required to cause argyria, all case reports to date are following excessive daily consumption of the element over a period of years10,11. Topical application of silver has been reported to cause localized argyria whereas systemic toxicity is generally the result of longstanding oral intake12. Argyria is more or less a benign condition characterized by a slate-grey metallic appearance of the skin. Apart from skin discoloration, extreme cases of systemic silver toxicity can be associated with thrombocytopenia, abnormal clotting, renal impairment, proteinuria, and neurological symptoms such as seizures, loss of coordination and sensory loss12. All of these possible side effects are exceedingly rare and are not expected to be an issue in this study. There is, however, a possibility that there might be localized pigmentation of the nasal mucosa, of which there are no significant consequences13.

Our goal with this project is to test whether topical silver colloid is a feasible treatment option for patients with refractory CRS. With the recent publication of a proof of mechanism study6, the investigators are looking to extend the same notion into a proof of concept investigation. The investigators propose taking twenty volunteer patients with recalcitrant CRS and trial randomized to a course of daily intranasal silver colloid for 6 weeks followed by saline, or vice versa. Pre and post-treatment measurements will be taken using validated scoring systems for CRS patients14-16. These include the Sino-Nasal Outcome Test (SNOT-22)14, Lund-Kennedy score15 and the Smell Identification Test16, which examine quality of life indices, endoscopic assessments and sense of smell, respectively. Should the results of this preliminary study be in favor of silver colloid use in CRS patients the investigator should look into arranging a formal Randomized-Controlled Clinical Trial.

ELIGIBILITY:
Inclusion Criteria:

* A history of twelve or more weeks with at least 2 of the following:

  * Nasal congestion
  * Mucus discharge from the nose or mucus that drips down the back of the throat
  * Facial pain or pressure
  * A decrease sense of smell
* A history of at least 2 of the following

  * One or more failed functional endoscopic sinus surgeries for CRS
  * Failed oral, culture-directed antibiotic therapy for CRS
  * Failed oral or topical steroid therapy for CRS
  * Failed baby shampoo nasal irrigation therapy for CRS
  * Failed topical mupirocin therapy for CRS
  * Failed Manuka honey irrigations for CRS
  * Failed budesonide irrigations for CRS

Exclusion Criteria:

* Patients with nasal polyposis
* Patients with existing autoimmune disorders
* Patients with an allergy to silver
* Patients with diabetes
* Patients that have previously used colloidal silver as a naturopathic remedy
* Patients that are pregnant, attempting/planning to become pregnant or breastfeeding
* Patients below the age of 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2015-12-10 (Actual); Primary Completion 2016-03-06 (Actual); Study Completion 2017-04-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leigh Sowerby, MD, Principal Investigator — Schulich School of Medicine and Dentistry/Otolaryngology
Locations (2):
- Canada (2):
  - Saint Joseph's Health Care, London, Ontario
  - St. Joseph's Health Care, London, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Scott JR, Krishnan R, Rotenberg BW, Sowerby LJ. The effectiveness of topical colloidal silver in recalcitrant chronic rhinosinusitis: a randomized crossover control trial. J Otolaryngol Head Neck Surg. 2017 Nov 25;46(1):64. doi: 10.1186/s40463-017-0241-z. PMID 29178954

RESULTS

PARTICIPANT FLOW:
Groups:
- Saline, Then Silver Colloid: Cross-over control Each participant does 6 weeks of topical nasal saline, followed by 6 weeks of topical nasal silver colloid (Dose= 6.7mcg silver daily; Frequency= 2 sprays in each nostril twice daily; Route= Topical intra-nasal spray; Duration= 6 weeks)
  Topical silver colloid: Patients will be provided with a standardized silver colloid spray and asked to place two sprays into each nostril twice daily for a total of 6 weeks. The commercially available silver colloid product, Sovereign Silver Mineral Supplement, will be used.
  Topical Saline
- Silver Colloid, Then Saline: Cross-over control Each participant receives 6 weeks of topical nasal silver colloid, followed by 6 weeks of saline (Dose= 6.7mcg silver daily; Frequency= 2 sprays in each nostril twice daily; Route= Topical intra-nasal spray; Duration= 6 weeks)
  Topical silver colloid: Patients will be provided with a standardized silver colloid spray and asked to place two sprays into each nostril twice daily for a total of 6 weeks. The commercially available silver colloid product, Sovereign Silver Mineral Supplement, will be used.
Period: Overall Study
Arm/Group | Saline, Then Silver Colloid | Silver Colloid, Then Saline
Started | 10 | 12
Completed | 8 | 12
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Saline Then Silver Colloid: Each participant uses 6 weeks of saline (Frequency= 2 sprays twice daily; Route= topical intra-nasal spray; Duration= 6 weeks) followed by 6 weeks of silver colloid (Dose= 6.7mcg silver daily; Frequency= 2 sprays twice daily; Route= Topical intra-nasal spray; Duration= 6 weeks)
- Silver Colloid Then Saline: Each participant uses 6 weeks of silver colloid (Dose= 6.7mcg silver daily; Frequency= 2 sprays twice daily; Route= Topical intra-nasal spray; Duration= 6 weeks) followed by 6 weeks of saline (Frequency= 2 sprays twice daily; Route= topical intra-nasal spray; Duration= 6 weeks).
- Total: Total of all reporting groups
Arm/Group | Saline Then Silver Colloid | Silver Colloid Then Saline | Total
Number analyzed (Participants) | 10 | 12 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 8 | 15
  >=65 years | 3 | 4 | 7
Age, Continuous [Mean (Full Range); unit: years] | 65.8 [44 to 86] | 62.3 [43 to 84] | 64.7 [43 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 2 | 8
  Male | 4 | 10 | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 10 | 12 | 22
SNOT-22 score [Mean (Standard Deviation); unit: units on a scale] — The SNOT-22 questionnaire is a 22-item document that assesses the social and emotional impact of CRS. Scores may range from 0-110 with higher scores representing more severe disease
  units on a scale | 59.3 (19.4) | 52.8 (19.2) | 54.2 (20.1)
Lund-Kennedy endoscopic score [Mean (Standard Deviation); unit: units on a scale] — The Lund Kennedy endoscopic score is an objective measure of the severity of CRS. Scores are given to reflect the degree of edema and obstruction within the various sinuses. Scores range from 0 to 12 with higher scores being worse.
  units on a scale | 7.8 (2.2) | 6.8 (2.3) | 7.1 (2.2)

OUTCOME MEASURES:

1. Primary Outcome: Change in Sino-nasal Outcome Test-22 Score Between Baseline and 6 Weeks, Then 6 Weeks to 12 Weeks.
Description: The Sinonasal Outcome Test-22 is a quality of life questionnaire examining the social and emotional distress of CRS. The scores range from 0 to 110 with higher scores representing more severe disease. Total score is reported. Higher values are a worse outcome.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Saline, Then Silver Colloid: Cross-over control Each participant does 6 weeks of topical nasal saline, followed by 6 weeks of topical nasal silver colloid (Dose= 6.7mcg silver daily; Frequency= 2 sprays in each nostril daily; Route= Topical intra-nasal spray; Duration= 3 months)
  Topical silver colloid: Patients will be provided with a standardized silver colloid spray and asked to place two sprays into each nostril daily for a total of three consecutive months. The commercially available silver colloid product, Sovereign Silver Mineral Supplement, will be used.
- Silver Colloid, Then Saline: Each participant receives the full 12 weeks of topical nasal silver colloid (Dose= 6.7mcg silver daily; Frequency= 2 sprays in each nostril daily; Route= Topical intra-nasal spray; Duration= 3 months)
  Topical silver colloid: Patients will be provided with a standardized silver colloid spray and asked to place two sprays into each nostril daily for a total of three consecutive months. The commercially available silver colloid product, Sovereign Silver Mineral Supplement, will be used.
Arm/Group | Saline, Then Silver Colloid | Silver Colloid, Then Saline
Number analyzed (Participants) | 8 | 12
units on a scale
  baseline | 59.3 (19.4) | 52.9 (19.2)
  6 weeks | 45.4 (16.8) | 51.8 (24.4)
  12 weeks | 49.3 (17.9) | 56.5 (23.5)

2. Primary Outcome: Change in Endoscopic Lund-Kennedy Score From Baseline to 6 Weeks, Then 6 Weeks to 12 Weeks
Description: Endoscopic evaluation of the individual paranasal sinuses (left and right) and the degree of obstruction of the osteomeatal unit. Scores range from 0 to 24 with a higher number representing more severe disease.
Time Frame: 6 weeks
Population: chronic rhinosinusitis without polyposis patients
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Saline Then Silver Colloid | Silver Colloid Then Saline
Number analyzed (Participants) | 8 | 12
score on a scale
  baseline | 7.8 (2.2) | 6.8 (2.3)
  6 weeks | 5.9 (1.6) | 5.7 (2.8)
  12 weeks | 4.8 (2.7) | 4.7 (1.6)

ADVERSE EVENTS:
Time Frame: Adverse events were collected over the entire 12 week period patients were enrolled in the study.
Groups:
- Saline Intervention: Adverse events that occurred during time using saline intervention are reported here.
- Colloidal Silver Intervention: Adverse events that occurred during time using colloidal silver intervention are reported here.
Arm/Group | Saline Intervention | Colloidal Silver Intervention
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 0/22 | 2/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Saline Intervention (N=22) | Colloidal Silver Intervention (N=22)
Acute exacerbation of sinusitis/severe nasal obstruction (Infections and infestations) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No